CLINICAL TRIAL: NCT02377024
Title: Effects of Tremella Fuciformis on Improvement in Cognitive-Bio-Markers of Cognitive Functions in Healthy Adults With Subjective Cognitive Impairment: An 8-Week Prospective Randomized Double-Blind Placebo-Controlled Trial With Multimodal Neuroimaging and Neurocognitive Assessments
Brief Title: Effects of Tremella Fuciformis on Improvement in Cognitive-Bio-Markers of Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBI_CT_TF
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Healthy Adults With Subjective Memory Complaints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- TF 600mg (Experimental): TF 600mg/day
  Interventions: Dietary Supplement: TF 600mg
- TF 1200mg (Experimental): TF 1200mg/day
  Interventions: Dietary Supplement: TF 1200mg
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: TF 600mg
  Arms: TF 600mg
Dietary Supplement: TF 1200mg
  Arms: TF 1200mg
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
The objective of this study is to demonstrate the cognitive enhancement effect and safety of Tremella Fuciformis, using the cognitive and clinical indicators (e.g. memory, attention, and psychomotor speed) and the latest brain imaging methods for healthy adults suffering subjective cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years old
* Global Deterioration Scale score (GDS) of 2
* High school or higher levels of education.

Exclusion Criteria:

* Current pregnancy or breast-feeding
* Evidence of neurologic or medical conditions
* Axis I diagnosis when assessed by the board certified psychiatrist using the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorder, 4th edition (DSM-IV)(SCID-IV)
* Mini-mental status examination score of 24 or less
* Clinical Dementia Rating score of 0.5 or more suggesting cognitive impairment beyond self-perceived subjective deficits
* Intelligence quotient less than 70
* Contraindications to magnetic resonance imaging (MRI)
* Use of psychotropics in last 3 months
* Use of oral contraceptive medication
* Participation in other clinical trials during the study period that might affect the outcome of the present study
* Allergic adverse reactions to mushrooms

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in neurocognitive function (neurocognitive test batteries such as CANTAB) | baseline, 8th week
  Scores from neurocognitive test batteries such as CANTAB
Changes from baseline in brain structure analyzed using the computational approach | baseline, 8th week
  Morphometric analysis of brain structures in magnetic resonance imaging
Changes from baseline in brain function analyzed using the computational approach (Blood oxygenation level dependent (BOLD) signal intensity) | baseline, 8 week
  Blood oxygenation level dependent (BOLD) signal intensity and their connectivity assessed using functional magnetic resonance imaging scans
Changes from baseline in brain biochemical metabolism analyzed using the computational approach (Brain metabolite concentrations assessed using magnetic resonance spectroscopy) | baseline, 8th week
  Brain metabolite concentrations assessed using magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Change from baseline in Subjective Memory Complaints Questionnaire scores at 8th weeks | baseline, 8th week
Number of participants with adverse events | 4th week
Number of participants with adverse events | 8th week

CONTACTS AND LOCATIONS:
Locations (1):
- Ewha Womans University, Seoul, South Korea